CLINICAL TRIAL: NCT07048054
Title: Allogenic Adipose-derived Stromal Cell Patch (i.e TrophiPatch, Provided by HekeTiss®) for Chronic Leg Ulcers Resistant to Standard Treatment: Safety and Preliminary Efficacy, a One-arm Monocentric Phase I-ll Trial
Brief Title: Safety and Preliminary Efficacy of TrophiPatch, an Adipose-Derived Stromal Cell Patch for Chronic Leg Ulcers
Acronym: RESCUE-PATCH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nicolò Brembilla (Other)
Responsible Party: Sponsor-Investigator, Nicolò Brembilla, Clinical study coordinator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00327
Record Dates: First submitted 2025-06-13; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot Ulcer (DFU); Venous Leg Ulcer (VLU)
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: One-arm monocentric phase I/lla trial of allogenic adipose-derived stromal cells for the treatment of chronic leg ulcers resistant to standard therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TrophiPatch treatment (Experimental): one time application of TrophiPatch
  Interventions: Drug: TrophiPatch: allogeneic adipose-derived stromal cell patch

INTERVENTIONS:
Drug: TrophiPatch: allogeneic adipose-derived stromal cell patch — Topical application of an allogeneic adipose-derived stromal cell patch

SUMMARY:
This study aims to evaluate the safety and effectiveness of an experimental biological dressing called TrophiPatch, applied to adults with chronic leg ulcers of diabetic or vascular orign. TrophiPatch contains stromal cells derived from a donor's fat tissue, which are purified and processed in a certified laboratory. These cells have shown wound-healing, anti-inflammatory and pro-angiogenic properties in preclinical studies.

All 18 participants will receive a single application of TrophiPatch on their wound. The total study duration is up to 24 weeks, with 23 scheduled visits for follow-up and monitoring.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older.
* Patients with more than one eligible ulcer will have one - usually the largest or more clinically significant - selected at screening as the index ulcer.
* Participants will have the capacity to understand study procedures, and will be able to providewritten informed consent.

(for VLU only)

* Diagnosed with at least one venous leg ulcer.
* Ulcers duration for 6 weeks to 3 years at the time of screening.
* Hard-to-healed ulcers with cross-sectional area that have decreased by less than 40% during a four-week run-in period.
* Reference ulcer surface from 5 to 25 cm2.
* At the time of inclusion, the ulcer will be clinically non-infected (TILI score ≥ 5).
* Absence of significant arterial insufficiency assessed at clinical examination (intermittent claudication or resting pain, necrotic or distal wound on the foot) and systolic homolateral ankle-brachial index (ABI) greater than 0.75 and inferior to 1.40 or biphasic or triphasic Doppler signals in the dorsalis or posterior tibial arteries of the affected limb.

(for DFU only)

* Patient with type 1 or type 2 diabetes.
* Diagnosed with at least one diabetic foot ulcer on a foot or both feet below the level of the malleoli, excluding ulcers confined to the interdigital cleft.
* Ulcers duration for 4 weeks to 3 years at the time of screening.
* Eligible ulcers will be hard-to-heal, meaning that the cross-sectional area will decrease by less than 50% during a four-week run-in period.
* Reference ulcer surface from 1 to 25 cm2.
* At the inclusion, the ulcer will be clinically non-infected (according to IDSA criteria).
* HbA1C < 12% at screening.
* Absence of significant arterial insufficiency assessed by systolic homolateral ankle-brachial index (ABI) greater than 0.75 and inferior to 1.40 or biphasic or triphasic Doppler signals in the dorsalis or posterior tibial arteries of the affected limb.

Exclusion Criteria

* Subject has a history of:

  * endstage renal disease
  * uncontrolled cardiac failure
  * severe malnutrition
  * severe liver disease
  * aplastic anemia
  * malignant disease (active or recent (<5 years))diabetes avec HbA1C > 12%
  * rheumatoid arthritis
  * sickle cell disease
  * other connective tissue disorder
  * irradiation to the affected extremity
* Serum creatinine concentration greater than 180 umol/L and/or receipt of renal dialysis or an estimated glomerular filtration rate (based on cystatin C or serum creatinine) of less than 20 mL/min per 1·73 m²
* Drug or alcohol abuse.
* Limited physical capacity or total immobility.
* Known pregnancy or nursing at the time of screening visit
* Subject is currently receiving (i.e within 30 days prior to inclusion) or scheduled to receive a medication or treatment that, in the opinion of the investigator, will interfere with or affect the rate of wound healing.
* Index ulcers probing to tendon, muscle, capsule and bone.
* Local or systemic signs of ongoing infection.
* Hypersensitivity to silicone or porcine gelatin.
* Previous treatment with growth factors, stem cells, or an equivalent preparation within the 8 weeks before the baseline visit.
* Involvement in another interventional clinical trial within the 4 weeks before the baseline visit.
* Known or suspected absence of capacity to understand the study procedures or provide written informed consent (decided by the investigator).
* Cross-sectional area of the index ulcer had increased by at least 20%.

(for VLU only)

* History of poor compliance with compression therapy.
* Presence of peripheral neuropathy of the lower limbs.

(for DFU only)

• History of poor compliance with offloading therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite safety outcome at week 12 from baseline | Week 12
  Composite outcome including any of the following events: deterioration of the ulcer, as measured by an increase of the ulcer size of > than 20% at week 12 as compared to d0; and/or presence of spreading infection or systemic infections (criteria according to IWII); and/or presence of treatment-related irritative or allergic contact dermatitis (as per clinical diagnosis)

SECONDARY OUTCOMES:
Number of patients with localised infection (TILI score ≥ 5) not suspicious for irritative or allergic contact dermatitis | Week 12
Extent of pruritus, as determined by Numerical Rating Score (NRS). | Week 12
  Eleven numbers from 0 to 10 are displayed and patients are asked to pick the number corresponding to the intensity of their pruritus
Number of patients with hyper-cicatrisation | Week 12
  Clinical evaluation
Number of patients with pathologic scar | Week 12
  clinical evaluation of cheloid or hypertrophic scar
Number of patients developing donor-HLA antibodies | Week 12
Weekly change in ulcer area till week 12 | from enrolment to week 12
  Standardised measurement of the wound area will be performed once weekly in the occasion of the first visit of the week using the SilhouetteTM camera. Change of wound area will be calculated by subtracting the surface area at week X to that measured at d0. This will be expressed as % of change with respect to d0.
Number of completely healed and epithelised ulcers at week 12. | Week 12
  Visual inspection of the ulcer at week 12 and evaluation of the corresponding digital image as acquired via the Silhouette camera. The ulcer will be considered completely healed if presenting an epithelial layer and persisting for 2 weeks.
Weekly evolution of the wound bed score till week 12 | From enrolment to week 12
  The wound bed score consists of 8 key components: (a) healing edges (wound edge effect); (b) black eschar; (c) greatest wound depth/granulation tissue; (d) amount of exudate, edema, peri-wound dermatitis, peri-wound callus and fibrosis; and (e) a pink wound bed. Each of these components is scored individually.. The maximum score (best score) is 16. The minimum possible score (worst score) is 0.
Evolution of the quality of blood perfusion of the wound | Week 2 and week 12
  The quality of vascularisation and the measurement of local oxygen (transcutaneous oximetry - tcpO2) will be determined by laser doppler imaging
Reduction in pain during the study period | From enrolment to week 12
  Pain will be measured using the Visual Analog Scale (VAS), a 10-centimeter horizontal line anchored by two extremes: "no pain" (score = 0) and "worst imaginable pain" (score = 10). Participants will indicate their pain level by marking a point on the line. Higher scores indicate worse pain.
Change in quality of life | Day 0 and week 12
  Change in quality of life will be assessed using the Wound-QoL questionnaire, a validated 17-item instrument specifically designed for patients with chronic wounds. Scores range from 0 to 4, with higher scores indicating worse quality of life.
Assessment of patient-relevant benefits during wound therapy | Day 0 and week 12
  Assessment of patient-relevant benefits during wound therapy will be conducted using the Patient Benefit Index (PBI), specifically the validated short version (PBI-S 2.0) and the PBI for chronic wounds (PBI-W). The PBI includes two parts: the Patient Needs Questionnaire (PNQ), where patients rate the importance of treatment goals, and the Patient Benefit Questionnaire (PBQ), where they rate the extent to which these goals were achieved. A weighted algorithm combines these ratings into a global PBI score ranging from 0 (no benefit) to 4 (maximum benefit). A score ≥ 1 is considered a clinically relevant benefit, while a score ≥ 3 reflects a high patient-reported benefit. Higher scores indicate greater perceived benefit from the therapy.

OTHER OUTCOMES:
Translational research - State of systemic and local (wound) inflammatory status | Enrolment, week 2 and 12
  Assessment of systemic and local inflammatory status using multiplex cytokine assays (e.g., Luminex) in plasma and wound fluid, as well as immunohistochemical staining for inflammatory markers in tissue sections.
Translational research - Persistence of TrophiPatch fibres and ASC cells | Enrolment, week 2 and 12
  Persistence of drug matrix fibers and adipose-derived stromal cells (ASCs) will be evaluated using histological staining (e.g., Masson's trichrome for matrix components and immunolabeling for ASC tracking).
Translational research - Development of anti-donor (HLA) specific antibodies | Enrolment, week 2 and 12
  Detection of anti-donor (HLA-specific) antibodies in serum using solid-phase assays such as Luminex Single Antigen Bead assays to monitor for humoral alloimmune responses.
Translational research - Local composition of the inflammatory infiltrate | enrolment, week 2 and 12.
  Characterization of the local inflammatory infiltrate within the healing wound by immunohistochemistry or immunofluorescence, targeting markers for resident and infiltrating cells: neutrophils, eosinophils, T cells, mast cells, macrophages, DCs.
Translational research - Local structure of dermal fibres within the healing wound | Enrolment, week 2 and 12
  Evaluation of dermal fiber structure and remodeling using routine histology and immunohistochemestry for collagen subtypes (e.g., Collagen I and III) and matrix proteins.
Translational research - Extent of Angiogenesis within the healing wound | Enrolment, week 2 and 12.
  Quantification of angiogenesis through immunohistochemical detection of endothelial markers (e.g., CD31, VEGF), along with image-based quantification of vessel density.
Translational research - Transcriptomic changes over time | Enrolment, week 2 and 12
  Transcriptomic profiling of wound tissue using bulk RNA sequencing (RNA-seq) or GeneChip arrays to analyze therapy-induced changes in gene expression over time.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland